CLINICAL TRIAL: NCT03648073
Title: [68Ga]DOTATATE-PET/MRI in Hepatocellular Carcinoma to Assess the Feasibility of Targeted Radionuclide Therapy With Somatostatin Receptor Ligands
Brief Title: [68Ga]DOTATATE-PET/MRI in Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Samuel Joseph Galgano, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R18-107
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Radiographic Evidence of HCC on CT or MRI (Experimental): [68Ga]DOTATATE-PET/MRI in Hepatocellular Carcinoma
  Interventions: Drug: [68Ga]DOTATATE-PET/MRI

INTERVENTIONS:
Drug: [68Ga]DOTATATE-PET/MRI — [68Ga]DOTATATE-PET/MRI

SUMMARY:
There is great need for new therapeutic options for patients with hepatocellular carcinoma (HCC). This proposal will assess the feasibility of a novel theranostic approach to HCC using [68Ga]DOTATATE, a recently approved positron emission tomography (PET) ligand for imaging somatostatin receptor (SSTR) positive tumors. In this study, we will use [68Ga]DOTATATE to determine the percentage of HCCs that express adequate levels of SSTR for treatment with targeted radionuclide therapy (TRT) using the therapeutic SSTR ligand [177Lu]DOTATATE. This radionuclide therapy was FDA approved in January 2018 for treating neuroendocrine tumors (NETs) arising from the gastrointestinal tract, but its use in HCC has not yet been explored. In the long term, we envision using [68Ga]DOTATATE-PET to identify HCC patients with adequate SSTR expression for TRT using [177Lu]DOTATATE.

Liver transplantation is the only curative therapy for HCC and is an option for a selected subset of HCC patients. For those who are not candidates for transplantation, locoregional therapies with limited efficacy are available such as percutaneous ablation, arterial chemoembolization, and Y-90 microsphere radionuclide therapies. There are few options for patients who progress or are not candidates for these therapies. The first line systemic therapy is sorafenib, a tyrosine kinase inhibitor. Sorafenib is often not well tolerated due to its side effects and there is need for additional systemic treatments. Multiple tissue-based studies demonstrate SSTR positivity in 20-50% of HCCs.[1-3] However, the fraction of HCCs have high enough levels of SSTR for [177Lu]DOTATATE therapy has not yet been assessed. This research plan is a critical prerequisite for determining the feasibility of this theranostic approach to treating HCC. If we obtain positive results, these data will be critical for designing a combined imaging and therapeutic study in HCC using DOTATATE.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of hepatocellular carcinoma, either by imaging criteria or pathology on biopsy
* Standard of care liver MRI or CT demonstrating viable HCC based on arterial contrast enhancement measuring at least 1.5 cm in largest axial dimension

Exclusion Criteria:

* History of neuroendocrine tumor or other SSTR-positive tumor
* Interval locoregional therapy or new systemic therapy between standard of care liver MRI or CT study showing viable HCC and [68Ga]DOTATATE-PET/MRI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Galgano, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Radiographic Evidence of HCC on CT or MR: [68Ga]DOTATATE-PET/MRI in Hepatocellular Carcinoma
  [68Ga]DOTATATE-PET/MRI: [68Ga]DOTATATE-PET/MRI
Period: Overall Study
Arm/Group | Patients With Radiographic Evidence of HCC on CT or MR
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Radiographic Evidence of HCC on CT or MR
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Demonstrating Somatostatin Receptor Positivity in Hepatocellular Carcinoma Using [68Ga]DOTATATE-PET
Time Frame: 1 PET/MRI scan
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Radiographic Evidence of HCC on CT or MR
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: During imaging study (including hour of uptake time and 90 minutes of imaging) and subsequent 24 hours post PET/MRI scan
Arm/Group | Patients With Radiographic Evidence of HCC on CT or MR
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT03648073/Prot_SAP_001.pdf